CLINICAL TRIAL: NCT00846196
Title: A Crossover Study to Assess the Bioequivalence of the Phase III and Commercial Risedronate 35 mg Delayed Release Formulations.
Brief Title: A Study to Assess the Bioequivalence of Different Formulations of Risedronate in Healthy Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 2008119
Record Dates: First submitted 2009-02-13; First posted 2009-02-18 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Risedronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Experimental): one commercial risedronate 35 mg DR tablet
  Interventions: Drug: risedronate 35 mg DR (Commercial Tablet)
- 1 (Active Comparator): one Phase III risedronate 35 mg DR tablet
  Interventions: Drug: risedronate DR (Phase III clinical supply)

INTERVENTIONS:
Drug: risedronate DR (Phase III clinical supply) — Reference - (Phase III clinical supply) one 35 mg DR tablet administered as a single oral dose after an overnight (10-hour) fast, followed by a 4-hour fast
  Other Names: Phase III clinical supply
  Arms: 1
Drug: risedronate 35 mg DR (Commercial Tablet) — Test - (Commercial tablets) one 35 mg DR tablet administered as a single oral dose after an overnight (10-hour) fast, followed by a 4-hour fast
  Other Names: Commercial Tablet
  Arms: 2

SUMMARY:
Randomized, double-blind, 2-treatment, 2-period, 2-sequence, crossover study, The study will consist of a screening visit, study center admission (preceding Treatment Periods 1 and 2), 2 treatment periods (4 days each), 1 washout period (14 to 17 days separating periods 1 and 2), and exit procedures.

ELIGIBILITY:
Inclusion Criteria:

* male or female, 18 to 65 years of age
* if female, non-lactating and either surgically sterile or postmenopausal
* body mass index less than or equal to 32 kg/m2 at screening

Exclusion Criteria:

* no use of a bisphosphonate within 1 month
* no history of GI disease
* no use of any medications within 7-14 days prior to scheduled dosing day

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 538 (Actual)
Dates: Start 2009-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Assess the bioequivalence (BE) between the commercial and the Phase III risedronate 35 mg DR formulations. | 72 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Chantell Wilson, PhD, Study Director — Procter and Gamble
Locations (6):
- United States (6):
  - Research Site, San Diego, California
  - Research Site, Fort Myers, Florida
  - Research Site, Miramar, Florida
  - Research Site, Omaha, Nebraska
  - Research site, Austin, Texas
  - Research Site, Dallas, Texas